CLINICAL TRIAL: NCT04016870
Title: Project My Heart Your Heart: Prospective Evaluation of the Safety and Efficacy of Cardiac Pacemaker Reuse in Low to Middle Income Countries
Brief Title: Project My Heart Your Heart: Pacemaker Reuse
Acronym: MHYH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Thomas Crawford, MD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00050238
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-04

CONDITIONS: Device Related Infection; Device Malfunction; Bradycardia
MeSH Terms: conditions — Prosthesis-Related Infections; Bradycardia

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, multi-center, single-blinded non-inferiority study of 278 patients (all outside of United States) with Class I indications for pacemaker implantation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- New Device (Active Comparator): New pacemakers will be sourced from pacemaker manufacturers.
  Interventions: Device: New Pacemaker
- Reconditioned Device (Experimental): Donated devices are inspected according to specific protocols that evaluate physical and electrical (battery longevity) suitability for future use. Devices deemed to be acceptable are shipped to a third-party vendor (NEScientific) for disassembly, cleaning and re-sterilization.
  Interventions: Device: Reconditioned Pacemaker

INTERVENTIONS:
Device: Reconditioned Pacemaker — Devices from the three manufacturers below will be used.
  Other Names: St. Jude Medical device; Boston Scientific device; Medtronic device
  Arms: Reconditioned Device
Device: New Pacemaker — Devices from the four manufacturers below will be used.
  Other Names: St. Jude Medical device; Boston Scientific device; Medtronic device; Biotronik device
  Arms: New Device

SUMMARY:
Lack of access to pacemakers is a major challenge to the provision of cardiovascular health care in Low and Middle Income Countries (LMIC). Post-mortem pacemaker utilization could be safe, efficacious, and ethically responsible means of delivering the needed care. Reconditioned pacemakers can provide therapy for patients with symptomatic bradycardia and no means of receiving a new device. The objective of the clinical trial is to determine if pacemaker reutilization can be shown to be a safe means of delivering pacemakers to patients in LMIC without resources. Consented patients in this multi-center trial will be randomized to undergo implantation of either a reconditioned device or a new device.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 2 years.
* Indications for device implantation must be fulfilled per standard of care. Consistent with 2008 American College of Cardiology / American Heart Association guidelines for device therapy, one of the following class I indications must be met.
* Sinus Node Dysfunction
* Acquired Atrioventricular (AV) Block
* Chronic Bifascicular Block
* Hypersensitive Carotid Syndrome
* Lack of financial ability to pay for a new device must be assessed and documented.
* All other methods of new device acquisition must be exhausted.
* Patient must be agreeable and able to follow-up with the implanting center within 2 weeks for wound check, at 2 months, 6 months, and every 6 months thereafter for routine pacemaker checks.

Exclusion Criteria:

* Severe valvular disease
* Severe pulmonary disease
* End-stage renal disease (creatinine clearance < 30 mL/min) whether or not on dialysis
* Evidence of ongoing systemic infection
* Prior pacemaker or implantable cardioverter-defibrillator implantation
* Significant contraindication to pacemaker implantation per evaluation of the implanting physician (very high risk of complications).
* Presence of any other condition that the local investigator feels would be problematic or would restrict or limit the participation of the patient for the entire study period
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2018-10-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Procedure-Related Infection at 12 months | 12 months post device implantation
  Clinical evidence of pacemaker infection includes local signs of inflammation at the generator site such as erythema, warmth, fluctuance, tenderness, purulent drainage, wound dehiscence, or erosion. Device related endocarditis will be reported if the Duke criteria for infective endocarditis are met. Procedure-related infections will be classified as follows: pocket infection, endocarditis, recurrent bacteremia, extrusion of wires or generator

SECONDARY OUTCOMES:
Freedom from Pacemaker Software or Hardware Malfunction at 12 months | 12 months post device implantation
  Pacemaker software or hardware malfunction include unexpected premature battery depletion, device or electrode malfunction, or unexplained patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Crawford, MD, Principal Investigator — University of Michigan
Locations (8):
- The Moi Teaching and Referral Hospital, Eldoret, Kenya
- Universidad Autonoma de Nuevo Leon, Monterrey, Mexico
- Hospital Central de Maputo, Maputo, Mozambique
- Nigeria (2):
  - LASUTH, Ikeja, Lagos
  - Port Harcourt Teaching Hospital, Port Harcourt, Rivers State
- FUNDACOR, Asunción, Paraguay
- Choithram Memorial Hospital, Freetown, Sierra Leone
- ASCARDIO, Barquisimeto, Lara, Venezuela

IPD SHARING:
Plan to Share IPD: No